CLINICAL TRIAL: NCT04766788
Title: Monitoring Beliefs and Physiological Measures in Students at Risk for COVID-19 Using Wearable Sensors and Smartphone Technology
Brief Title: Studying Students at Risk for COVID-19
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Sung Won Choi, Edith S Briskin and Shirley K Schlafer Foundation Research Professor of Pediatrics and Associate Professor of Pediatrics and Communicable Diseases, University of Michigan
Other Study IDs: HUM00185391
Record Dates: First submitted 2021-02-22; First posted 2021-02-23 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Covid19
Keywords: Wearable Sensors, students
MeSH Terms: conditions — COVID-19 | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Wearable devices, saliva samples, survey measures — Provide a self-collected saliva sample, download and use the suite of apps (e.g., Fitbit, Social Rhythms, Roadmap 2.0), and answer online surveys.

SUMMARY:
The goal of this longitudinal observational study is to learn about how the COVID-19 has impacted and continues to impact students at the University of Michigan. We hope to determine whether a combination of (1) continuous heart rate obtained from wearable devices, (2) self-reported data from surveys and symptom logs, and (3) saliva samples can be used to help students self-monitor for infection and eventually be able to create a predictive model to detect illness early.

DETAILED DESCRIPTION:
The study was originally intended to last one year, however, it was expanded to follow the study participants over several years.

During this study, participants will be asked to:

* Provide a baseline self-collected saliva sample
* Download and use a suite of mobile apps (e.g., Fitbit, Social Rhythms, Roadmap 2.0)
* Complete surveys online
* Wear non-invasive Fitbit smartwatch
* Grant the study team access to their university academic records (optional)

The study will use these tools to monitor participants' physical activity and mental health over the course of at least three years. The study will also examine whether there is a connection between mental health and academic performance.

ELIGIBILITY:
Inclusion Criteria:

* Students at the University of Michigan who have moved back to Ann Arbor or who are completing schooling completely online.
* For those completing school online, must be able to provide a mailing address within the United States where they can receive study tools
* Possession of a smartphone (Apple or Andriod)
* Ability to understand and demonstrate willingness to sign a written informed consent.

Exclusion Criteria:

* Unwilling or unable to comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students at the University of Michigan must be either coming to campus or reside in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 2381 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of wearing Fitbit device | 4 months
  Feasibility will will be defined as wearing the Fitbit watch at least 8 hours per day up to at least 5 days of the week

SECONDARY OUTCOMES:
Survey completion | Up to 9 months
  Completion will be measured by the number of participants who complete the study surveys
Saliva sample | Up to 4 months
  Analyze samples to determine a possible early prediction/detection model for COVID-19
Continuous heart rate | Up to 8 months
  Analyze heart rate data to determine a possible early prediction/detection model for COVID-19
Mental well-being | Up to 9 months
  Assess participant mental well-being during the COVID-19 pandemic and if the use of health and well-being applications impacts self-rated well-being

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Choi, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cislo C, Clingan C, Gilley K, Rozwadowski M, Gainsburg I, Bradley C, Barabas J, Sandford E, Olesnavich M, Tyler J, Mayer C, DeMoss M, Flora C, Forger DB, Cunningham JL, Tewari M, Choi SW. Monitoring beliefs and physiological measures in students at risk for COVID-19 using wearable sensors and smartphone technology: Protocol for a mobile health study. JMIR Res Protoc. 2021 Jun 4;10(6):e29561. doi: 10.2196/29561. Online ahead of print. PMID 34115607
- [Background] Gilley KN, Baroudi L, Yu M, Gainsburg I, Reddy N, Bradley C, Cislo C, Rozwadowski ML, Clingan CA, DeMoss MS, Churay T, Birditt K, Colabianchi N, Chowdhury M, Forger D, Gagnier J, Zernicke RF, Cunningham JL, Cain SM, Tewari M, Choi SW. Risk Factors for COVID-19 in College Students Identified by Physical, Mental, and Social Health Reported During the Fall 2020 Semester: Observational Study Using the Roadmap App and Fitbit Wearable Sensors. JMIR Ment Health. 2022 Feb 10;9(2):e34645. doi: 10.2196/34645. PMID 34992051
- [Derived] Jayaraj G, Cao X, Horwitz A, Rozwadowski M, Shea S, Hanauer SN, Hanauer DA, Tewari M, Shedden K, Choi SW. Trends in Mental Health Outcomes of College Students Amid the Pandemic (Roadmap mHealth App): Longitudinal Observational Study. J Med Internet Res. 2025 Jan 9;27:e67627. doi: 10.2196/67627. PMID 39787592